CLINICAL TRIAL: NCT01872494
Title: Pain Treatment in Posterior Thoracolumbar Operation a Randomized Study to Assess the Effect of Local Analgesia After Operation
Brief Title: The Impact of Local Analgesia for Postoperative Analgesia in Posterior Thoracolumbar Operation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: local anaesthetic
Record Dates: First submitted 2013-05-24; First posted 2013-06-07 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: Local analgesia system; Ropivacaine; Analgesic efficacy after operation; Postoperative
MeSH Terms: conditions — Pain | interventions — Ropivacaine; flurbiprofen axetil; Palonosetron; Pentazocine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local (Experimental): This group uses local analgesia infusion pump of 0.33% ropivacaine 250ml through the wound for postoperative analgesia.
  Interventions: Other: local; Drug: 0.33% ropivacaine 250ml
- intravenous (Active Comparator): This group is treated with intravenous analgesia pump infusion of flurbiprofen axetil 150mg,palonosetron 0.5mg,pentazocine 240mg.
  Interventions: Other: intravenous; Drug: flurbiprofen axetil 150mg,palonosetron 0.5mg,pentazocine 240mg.

INTERVENTIONS:
Other: local — This group uses local analgesia infusion pump of 0.33% ropivacaine 250ml through the wound for postoperative analgesia.
  Arms: Local
Other: intravenous — This group is treated with intravenous analgesia pump infusion of flurbiprofen axetil 150mg,palonosetron 0.5mg,pentazocine 240mg.
  Arms: intravenous
Drug: 0.33% ropivacaine 250ml
  Arms: Local
Drug: flurbiprofen axetil 150mg,palonosetron 0.5mg,pentazocine 240mg.
  Arms: intravenous

SUMMARY:
Posterior thoracolumbar operation always chooses general anesthesia. Due to surgical trauma and rich periosteum and joint capsule innervation, patients after general anesthesia immediately feel acute pain.The use of appropriate postoperative analgesia in patients with thoracolumbar surgery is beneficial to postoperative recovery. Infusions of local anaesthetic via multilumen catheters that deliver directly to wound sites have been used for postoperative analgesia in procedures. Reducing the morbidity from both pain and nausea will make the mode of analgesia a better tolerated and more palatable option for patients. The aim of this study is to examine the effects of using local anaesthetic infusion catheters following posterior thoracolumbar surgery, and compares the outcomes of patients managed using intravenous analgesia pump infusion of systemic opioids.

DETAILED DESCRIPTION:
All 71 adult patients were prospectively included and randomized to either the local (L) group (n=35) or the intravenous (V) group (n=36) by using a random number table: the test group were treated with local analgesia infusion pump of 0.33% ropivacaine through the wound for postoperative analgesia, while the control group were treated with intravenous analgesia pump infusion of flurbiprofen axetil,palonosetron, pentazocine. At 2, 4, 6, 12, 24, 36, 48 hours after operation, postoperative pain visual analogue scale(VAS) scores and sedation Ramsay scores were used to evaluate the level of pain and sedation, and investigators documented the comprehensive evaluation of patients with pain control system, and the incidence of adverse reactions. At 24, 48 hours investigators observed the wound whether inflammation and exudation or not, and the removal of penetration catheter sent to clinical laboratory for bacterial culture. Investigators also recorded the length of time to discharge and called to ask pain conditions at the first 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ patient undergoing elective posterior thoracolumbar operation
2. between 18 and 70 years of age

Exclusion Criteria:

1. A history of cardiopulmonary disease, liver and kidney dysfunction, abnormal coagulation
2. Preoperative use of analgesic drugs
3. A allergy history of ropivacaine and polyurethane material

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
pain | 48 hours postoperation
  Up to 48 hours after operation,postoperative pain visual analogue scale(VAS) scores are used to evaluate the level of pain.

SECONDARY OUTCOMES:
sedation | 48 hours postoperation
  At 2, 4, 6, 12, 24, 36, 48 hours after operation,sedation Ramsay scores are used to evaluate the level of sedation.
comprehensive evaluation | 48 hours postoperation
  Investigators document the comprehensive evaluation of patients with pain control system,including the incidence of adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jirarattanaphochai K, Jung S, Thienthong S, Krisanaprakornkit W, Sumananont C. Peridural methylprednisolone and wound infiltration with bupivacaine for postoperative pain control after posterior lumbar spine surgery: a randomized double-blinded placebo-controlled trial. Spine (Phila Pa 1976). 2007 Mar 15;32(6):609-16; discussion 617. doi: 10.1097/01.brs.0000257541.91728.a1. PMID 17413463
- [Background] Mekawy N M, Badawy S S I, Sakr S A. Role of postoperative continuous subfascial bupivacaine infusion after posterior cervical laminectomy: Randomized control study. Egyptian J Anaesth, 2012, 28(1): 83-88.
- [Background] Aguirre J, Baulig B, Dora C, Ekatodramis G, Votta-Velis G, Ruland P, Borgeat A. Continuous epicapsular ropivacaine 0.3% infusion after minimally invasive hip arthroplasty: a prospective, randomized, double-blinded, placebo-controlled study comparing continuous wound infusion with morphine patient-controlled analgesia. Anesth Analg. 2012 Feb;114(2):456-61. doi: 10.1213/ANE.0b013e318239dc64. Epub 2011 Nov 10. PMID 22075018